CLINICAL TRIAL: NCT05666375
Title: Percutaneous Translumbar Vs Transhepatic Insertion of Long Term Hemodialysis Catheters (Permcath) After Failure of Classic Accesses
Brief Title: Percutaneous Translumbar Vs Transhepatic Permcath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Morsy Mohamed Khalil, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Unconventional permcath
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous translumbar permcath (Active Comparator): * Local anesthesia in adults and general anesthesia in pediatrics.
  * The patient under fasting condition is placed prone on angiography table.
  * Skin preparation and a sterile draping of the operating field.
  * Puncture site is chosen 1.5 cm above right iliac crest 10 cm lateral to the posterior median line.
  * Puncture into inferior vena cava is made using 21 gauge 15 cm long needle, inserted at 45 degree angle from the horizontal and advanced medially and superiorly under us then fluoroscopic guidance.
  * Entry into the IVC is made below the level of the renal veins, immediately anterior to the 3rd lumber vertebra.
  * Intravascular position of the needle is confirmed by free aspiration of blood and injection of contrast media under fluoroscopy.
  * A guide wire is introduced through the needle and advanced well into the IVC.
  * The needle is replaced with a dilator. A catheter of appropriate length is tunneled subcutaneously from the right flank and advanced to the IVC
  Interventions: Procedure: Percutaneous translumbar and transhepatic permcath
- Percutaneous transhepatic permcath (Active Comparator): * The patient lies in supine position.
  * The procedure is done under local anesthesia.
  * Under ultrasound guidance; access by a 21 gauge angiocatheter (15cm) to right or middle hepatic vein through intercostal or subcostal approach.
  * Entrance of the hepatic veins is confirmed by injection of diluted contrast media (iopromide) under fluoroscopy.
  * A 0.018-inch guidewire is advanced through the needle and into the right atrium.
  Intravascular catheter length is measured and selected in standard fashion.
  * The initial access needle is exchanged over the guidewire for a coaxial transitional sheath, which permits replacement of the 0.018-inch guidewire with a 0.035-inch guidewire.
  * The tunneled catheter is inserted over the wire through a peel-away sheath
  Interventions: Procedure: Percutaneous translumbar and transhepatic permcath

INTERVENTIONS:
Procedure: Percutaneous translumbar and transhepatic permcath — For selected ESRD patients who have exhausted all conventional access routes , translumbar and transhepatic insertion of long term hemodialysis catheters provide additional sites for access

SUMMARY:
The aim of the study is to emphasize the technique , success rate , efficacy of translumbar and transhepatic approaches and shed light on the complications of both methods and through comparison we can give recommendations to either of these methods.

DETAILED DESCRIPTION:
For selected ESRD patients who have exhausted all conventional access routes , translumbar and transhepatic permcath provide additional sites for access. This study will compare the two methods in terms of technical success (position of catheter tip), patency (primary defined as the number of catheter days from initial placement until removal & secondary defined as the number of catheter days after device replacement using the same access site) , mean cumulative duration of catheter in situ defined as the cumulative catheter days divided by the number of patients, function (adequacy of dialysis based on Urea Reduction Ratio URR & Simplified Daugirdas Formula Kt/V) and complications (infectious; exit site infection & sepsis and non-infectious; thrombosis, catheter migration, hematoma, intraperitoneal hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

- Chronic dialysis patients with failed classic routes of catheterization ( internal jugular, subclavian and femoral veins bilaterally ) as well as non-functioning a-v fistulas.

Exclusion Criteria:

1. Patients with uncorrectable coagulopathy.
2. Patients on long term anticoagulants
3. Concurrent active infection.
4. Sgnificant abdominal ascites. (transhepatic)
5. Cirrhotic liver disease patients. (transhepatic)
6. Morbid obesity. (translumbar)

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Catheter patency | Baseline
  patency (primary defined as the number of catheter days from initial placement until removal & secondary defined as the number of catheter days after device replacement using the same access site) , mean cumulative duration of catheter in situ defined as the cumulative catheter days divided by the number of patients

REFERENCES:
- [Background] Kade G, Les J, Buczkowska M, Labus M, Niemczyk S, Wankowicz Z. Percutaneous translumbar catheterization of the inferior vena cava as an emergency access for hemodialysis - 5 years of experience. J Vasc Access. 2014 Jul-Aug;15(4):306-10. doi: 10.5301/jva.5000185. Epub 2013 Nov 4. PMID 24190069
- [Background] Lorenz JM. Unconventional venous access techniques. Semin Intervent Radiol. 2006 Sep;23(3):279-86. doi: 10.1055/s-2006-948767. PMID 21326774
- [Background] Napalkov P, Felici DM, Chu LK, Jacobs JR, Begelman SM. Incidence of catheter-related complications in patients with central venous or hemodialysis catheters: a health care claims database analysis. BMC Cardiovasc Disord. 2013 Oct 16;13:86. doi: 10.1186/1471-2261-13-86. PMID 24131509
- [Background] Farag YMK, El-Sayed E. Global Dialysis Perspective: Egypt. Kidney360. 2022 Apr 20;3(7):1263-1268. doi: 10.34067/KID.0007482021. eCollection 2022 Jul 28. No abstract available. PMID 35919518
- [Background] Zouaghi MK, Lammouchi MA, Hassan M, Rais L, Krid M, Smaoui W, Jebali H, Kheder R, Hamida FB, Moussa FB, Fatma LB, Beji S. Determinants of patency of arteriovenous fistula in hemodialysis patients. Saudi J Kidney Dis Transpl. 2018 May-Jun;29(3):615-622. doi: 10.4103/1319-2442.235183. PMID 29970738